CLINICAL TRIAL: NCT00478010
Title: Research Participation: Decision Making and Outcomes in Cancer Clinical Trials
Brief Title: Making Decisions About Participating in a Cancer Clinical Trial for Patients With Stage II, Stage III, or Stage IV Pancreatic Cancer or Stage III or Stage IV Colon Cancer or Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Health Services Research
Other Study IDs: J0666; P30CA006973 (NIH); JHOC-J0666; CDR0000530879; NA_00003458 (Other: JHM IRB)
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2010-08

CONDITIONS: Colorectal Cancer; Pancreatic Cancer; Psychosocial Effects of Cancer and Its Treatment
Keywords: psychosocial effects of cancer and its treatment; stage III colon cancer; stage IV colon cancer; stage III rectal cancer; stage IV rectal cancer; stage II pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Counseling; Psychiatric Rehabilitation

INTERVENTIONS:
Other: counseling intervention
Other: study of socioeconomic and demographic variables
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Determining how patients makes decisions about participating in a clinical trial may help doctors plan clinical trials in which more patients are willing to participate and are satisfied with their decision to participate.

PURPOSE: This clinical trial is studying how patients with stage II, stage III, or stage IV pancreatic cancer or stage III or stage IV colon cancer or rectal cancer make decisions about participating in a clinical trial.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the relationship between disease factors, patient factors, and understanding of the cancer clinical trial, and preferences for decision control in the decision to participate in a cancer clinical trial by patients with stage II-IV pancreatic cancer or stage III-IV colon or rectal cancer.
* Determine the relationship between disease factors, patient factors, understanding of the cancer clinical trial, and preferences for decision control with satisfaction with the decision to participate in a cancer clinical trial.
* Determine how quality of life, trust, and hope impact the decision to participate in a cancer clinical trial and the satisfaction with this decision.

OUTLINE: This is a cross-sectional study.

Patients complete 12 questionnaires to assess their symptom burden (e.g., nausea, pain, fatigue), sociodemographics, hope, quality of life, trust in the healthcare system, trust in health professionals, research decision control, perceived risks, adequacy of research information, clinical trial participation, and decision satisfaction.

PROJECTED ACCRUAL: A total of 200 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Stage II-IV pancreatic cancer
  * Stage III-IV colon cancer
  * Stage III-IV rectal cancer
* Offered the opportunity to participate in a phase I-III cancer clinical trial and agreed or declined to participate
* First appointment at the Sidney Kimmel Comprehensive Cancer Center at John Hopkins

PATIENT CHARACTERISTICS:

* Able to read English

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2007-01-19 (Actual); Primary Completion 2008-09-29 (Actual); Study Completion 2008-09-29 (Actual)

PRIMARY OUTCOMES:
Participation
Decision satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Biedrzycki, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States